CLINICAL TRIAL: NCT00466778
Title: Autonomic Nervous System Dysfunction and Peripheral Neuropathy in a Cohort of Asymptomatic Juvenile Diabetic Patients (Type I): A Case-Controlled Study
Status: Completed | Type: Observational
Sponsor: Weintraub, Michael I., MD, FACP, FAAN (Individual)
Other Study IDs: 2007425
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Peripheral Neuropathy; Autonomic Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a case-controlled study using an innovative, non-invasive, FDA approved technology to measure the autonomic nervous system. Detection of unsuspected DPN or ANS dysfunction may allow physicians to re-assess current treatment and develop new dietary or pharmacological strategies. This also is an immense public health concern since there are currently 18 million diabetics in the United States and 220 million worldwide.

DETAILED DESCRIPTION:
A consecutive cohort of 20 neurologically asymptomatic (absence of numbness, tingling, burning or pain in the feet) patients with Type I from the practice of Dr. Richard Noto (gatekeeper) and associates will be asked with their legal guardians to enroll in this case-controlled study using a battery of safe, neurological tests which are unlikely to be painful. A second group of 20 subjects who are nondiabetic and healthy (age/sex matched) will also be enrolled and undergo the same battery of neurological tests. The battery of tests is highly accurate, objective and safe. Subjects will be referred and enrolled from the private practices of community pediatricians. A BMI derived from the subject's height and weight will be assessed by Dr. Noto. Subjects who are felt to be acceptable by the inclusion criteria will then receive consecutive numbers from 1 to 40 and their initials will follow their specific number for each study.

ELIGIBILITY:
Inclusion Criteria:

* Cooperation of the subject and guardian are required for this 60-120 minute evaluation.
* Capable of understanding and complying with study protocol.
* Twenty (20) male/females with juvenile diabetes [of at least 3 years duration and no longer than 7] (Type I) who are neurologically asymptomatic without numbness, tingling, burning or pain in the feet, ages 10-18.
* Fasting blood glucose greater than 120 mg at the time of initial diagnosis or a HbA1C greater than 6.0 at the time of the initial diagnosis will indicate that individual is to be considered a diabetic.
* BMI ranges of acceptability are greater than 5th percentile and less than 85th percentile.

Exclusion Criteria:

* Symptomatic with neurological symptoms of numbness, tingling, burning or pain in the feet of either controls or diabetic subjects.
* On medications that can produce peripheral neuropathy, i.e. statins (Lipitor), Dilantin, anti-neoplastic drugs.
* Unable to understand informed consent, i.e. mental retardation, psychosis, communicative impairment, language barrier.
* Morbid obesity - maximum BMI greater than 85th percentile.
* Underweight status less than 5th percentile BMI.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Noto, MD, Study Chair — Phelps Memorial Hospital
Locations (1):
- Michael I. Weintraub, MD, Briarcliff Manor, New York, United States